CLINICAL TRIAL: NCT00047593
Title: Phase 3 Study to Compare Two Different IOP Lowering Medications for the Treatment of Open Angle Glaucoma or Ocular Hypertension in Japanese Subjects C-01-98.
Brief Title: Phase 3 Study Comparing IOP Lowering in OAG or OH in Japanese Subjects C-01-98
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-01-98; C-01-98
Record Dates: First submitted 2002-10-08; First posted 2002-10-11 (Estimated); Last update posted 2008-08-05 (Estimated); Status verified 2008-08

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
Keywords: open-angle; glaucoma; ocular; hypertension; POAG; Iris; Pigmentation; Japanese
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma; Hypertension

INTERVENTIONS:
Drug: IOP Lowering Medications

SUMMARY:
The purpose of this study is to evaluate safety and efficacy of two different IOP lowering medications after twelve months of treatment in Japanese subjects.

ELIGIBILITY:
Adults of Japanese Ethnicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-01; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Los Angeles, California
  - San Francisco, California
  - Honolulu, Hawaii